CLINICAL TRIAL: NCT02686723
Title: Evaluation of Clinical and Biomechanical Correlation During Return to Sport After Anterior Cruciate Ligament Injury
Acronym: REPILOG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RB15.162
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-01

CONDITIONS: ACL Injury
Keywords: ACL injury; Return to sport; Motion analysis; Isokinetic evaluation; Risk factor
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACL injury (Experimental): Subjects who has ACL injury repaired and who were allowed to return to sport
  Interventions: Other: Clinical and biomechanical evaluations
- Healthy subjects (Active Comparator): Subjects who has never been injured in ACL and who practice sports with cutting task (soccer, handball)
  Interventions: Other: Clinical and biomechanical evaluations

INTERVENTIONS:
Other: Clinical and biomechanical evaluations — Clinical evaluation : demographics, clinic and functional testing. Biomechanical evaluation : isokinetic, motion analysis of 2 specific motion (drop vertical jump and cutting task) and anterior tibial translation with GnRB

SUMMARY:
Comparison of two groups of subjets (ACL injury who return to sport) and control group non-injured about clinical and biomechanical data :

* clinical test
* functional test
* motion analysis of 2 sport exercises
* tibial translation
* isokinetic evaluation

DETAILED DESCRIPTION:
ACL injury in sport practice is frequent and after surgery subjects want to return to sport. Re injury during return to sport is significant and clinical and biomechanical risk factors are described. But no study investigate link between clinical and biomechanical during this risk period.

The study will search to highlight correlation between clinical and biomechanical factors. Investigators will realize clinical evaluation (pain, translation) and functional tests (single hop test, triple hop test, 6m time hop test, crossover test). For biomechanical data, investigators will test 2 exercises in motion analyse laboratory (drop vertical jump and cutting task), a translation knee test with GnRB and isokinetic evaluation.

Investigators will compared results of injured subjects with a control group non-injured.

ELIGIBILITY:
Inclusion Criteria:

* surgeon repair ACL injury ; sport practice ; signed informed consent

Exclusion Criteria:

* for injury subjects: pain during cutting tasks ; associated injury with ACL rupture
* for healthy subjects: history of ACL injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Limb Symmetry Index | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REMY-NERIS, MD, PhD, Principal Investigator — University Hospital Brest, France
Locations (1):
- University Hospital, Brest, France

REFERENCES:
- [Background] Granan LP, Bahr R, Steindal K, Furnes O, Engebretsen L. Development of a national cruciate ligament surgery registry: the Norwegian National Knee Ligament Registry. Am J Sports Med. 2008 Feb;36(2):308-15. doi: 10.1177/0363546507308939. Epub 2007 Nov 7. PMID 17989167
- [Background] Olsen OE, Myklebust G, Engebretsen L, Bahr R. Injury mechanisms for anterior cruciate ligament injuries in team handball: a systematic video analysis. Am J Sports Med. 2004 Jun;32(4):1002-12. doi: 10.1177/0363546503261724. PMID 15150050
- [Background] Herbst E, Hoser C, Hildebrandt C, Raschner C, Hepperger C, Pointner H, Fink C. Functional assessments for decision-making regarding return to sports following ACL reconstruction. Part II: clinical application of a new test battery. Knee Surg Sports Traumatol Arthrosc. 2015 May;23(5):1283-1291. doi: 10.1007/s00167-015-3546-3. Epub 2015 Feb 28. PMID 25724802
- [Background] Crawford SN, Waterman BR, Lubowitz JH. Long-term failure of anterior cruciate ligament reconstruction. Arthroscopy. 2013 Sep;29(9):1566-71. doi: 10.1016/j.arthro.2013.04.014. Epub 2013 Jun 29. PMID 23820260
- [Background] Webster KE, Feller JA, Leigh WB, Richmond AK. Younger patients are at increased risk for graft rupture and contralateral injury after anterior cruciate ligament reconstruction. Am J Sports Med. 2014 Mar;42(3):641-7. doi: 10.1177/0363546513517540. Epub 2014 Jan 22. PMID 24451111
- [Background] Ford KR, Myer GD, Hewett TE. Valgus knee motion during landing in high school female and male basketball players. Med Sci Sports Exerc. 2003 Oct;35(10):1745-50. doi: 10.1249/01.MSS.0000089346.85744.D9. PMID 14523314
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287
- [Background] Paterno MV, Schmitt LC, Ford KR, Rauh MJ, Myer GD, Huang B, Hewett TE. Biomechanical measures during landing and postural stability predict second anterior cruciate ligament injury after anterior cruciate ligament reconstruction and return to sport. Am J Sports Med. 2010 Oct;38(10):1968-78. doi: 10.1177/0363546510376053. Epub 2010 Aug 11. PMID 20702858